CLINICAL TRIAL: NCT00727272
Title: A Relative Bioavailability Study of Quinine Sulfate Capsules Under Fasting and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Matthew Davis, MD, Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RA3-085
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2009-12-30 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Bioavailability
MeSH Terms: interventions — Quinine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Quinine Sulfate Caps 324 mg - Fasting (Experimental): A single dose of quinine sulfate 324 mg administered with 240 mL of room temperature water after an overnight fast of at least 10 hours.
  Interventions: Drug: Quinine Sulfate Capsules 324 mg
- Quinine Sulphate Tabs 300 mg - Fasting (Experimental): A single dose of quinine sulphate 300 mg administered with 240 mL of room temperature water after an overnight fast of at least 10 hours.
  Interventions: Drug: Quinine Sulphate Tablets 300 mg
- Quinine Sulfate Caps 324 mg - Fed (Experimental): A single dose of quinine sulfate 324 mg administered with 240 mL of room temperature water thirty minutes after the initiation of a standardized, high-fat breakfast.
  Interventions: Drug: Quinine Sulfate Capsules 324 mg

INTERVENTIONS:
Drug: Quinine Sulfate Capsules 324 mg — One 324 mg capsule administered after an overnight fast of at least 10 hours.
  Arms: Quinine Sulfate Caps 324 mg - Fasting
Drug: Quinine Sulphate Tablets 300 mg — One 300 mg tablet administered after an overnight fast of at least 10 hours.
  Arms: Quinine Sulphate Tabs 300 mg - Fasting
Drug: Quinine Sulfate Capsules 324 mg — One 324 mg capsule administered thirty minutes after the initiation of a standardized, high-fat breakfast.
  Arms: Quinine Sulfate Caps 324 mg - Fed

SUMMARY:
The purpose of this study is to evaluate and compare the relative bioavailability of Quinine Sulfate 324 mg capsules, manufactured by the Mutual Pharmaceutical Company, to Quinine Sulphate 300 mg tablets, manufactured by the Government Pharmaceutical Organization, Bangkok Metropolis, Thailand, after single oral dose administration under fasting conditions. An additional purpose of this study is to evaluate the effect of food on the Mutual Pharmaceutical Company product.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and compare the relative bioavailability of Quinine Sulfate 324 mg capsules, manufactured by the Mutual Pharmaceutical Company, to Quinine Sulphate 300 mg tablets, manufactured by the Government Pharmaceutical Organization, Bangkok Metropolis, Thailand, after single oral dose administration under fasting conditions. An additional purpose of this study is to evaluate the effect of food on the Mutual Pharmaceutical Company product.

Twenty-seven healthy, non-smoking, non-obese, male and female volunteers at least 18 years of age will be randomly assigned in crossover fashion to receive each of three dosing regimens in sequence with a 7 day washout period between dosing periods. In each of the three dosing periods, after a fast of at least 10 hours, subjects will receive one dose of one of the three test products (treatment A - quinine sulfate capsules 324 mg, treatment B - quinine sulphate tablets 300 mg, treatment C - quinine sulfate capsules 324 mg administered thirty minutes after the initiation of a standardized, high-fat breakfast). Subjects will fast for 4 hours after dosing. Blood samples will be drawn from all participants before dosing and for 48 hours post-dose at times sufficient to adequately define the pharmacokinetics of quinine sulfate under fed and fasting conditions and quinine sulphate under fasting conditions. Sitting blood pressure and heart rate will be obtained prior to dosing and at 1, 2, 4 and 12 hours post-dose and upon completion of the study. An electrocardiogram will be recorded at check-in and at 2, 4, 6, 12, and 24 hours post-dose. Subjects will be monitored throughout their participation in the study for adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All volunteers selected for this study will be healthy men or women at least 18 years of age, inclusive, at the the time of dosing. The weight range will not exceed ± 20% for height and body frame as per Desirable Weights for Adults - 1983 Metropolitan Height and Weight Table
* Screening procedures: Each volunteer will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.
* Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.
* The screening clinical laboratory procedures will include:
* HEMATOLOGY: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count
* CLINICAL CHEMISTRY:serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase
* HIV antibody and hepatitis B surface antigen screens
* URINALYSIS: by dipstick; full microscopic examination if dipstick positive; and
* URINE DRUG SCREEN: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine
* SERUM PREGNANCY SCREEN (female volunteers only)

If female and:

* of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condom with spermicide, diaphragm, intrauterine device (IUD), or abstinence; or
* is postmenopausal for at least 2 years; or
* is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators)
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant
* Volunteers demonstrating a positive hepatitis B surface antigen screen or a reactive HIV antibody screen
* Volunteers demonstrating a positive drug screen when screened for this study
* Female volunteers demonstrating a positive pregnancy screen
* Female volunteers who are currently breastfeeding
* Volunteers with a history of allergic response(s) to quinine or related drugs
* Volunteers with a history of clinically significant allergies including drug allergies
* Volunteers with a history of clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators)
* Volunteers who currently use tobacco products
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing
* Volunteers who report donating greater than 150mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study
* Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study
* Volunteers who report receiving any investigational drug within 28 days prior to Period I dosing
* Volunteers who report taking any systemic prescription medication in the 14 days prior to Period I dosing
* Volunteers with QTc >480 msec on the screening electrocardiogram (ECG) or with clinically significant findings
* Volunteers who have a glucose-6-phosphate dehydrogenese deficiency (G6PD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-02; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm.D., Principal Investigator — PRACS
Locations (1):
- PRACS, Fargo, North Dakota, United States

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence ABC; Treatment Sequence BCA; Treatment Sequence CAB: All subjects received each of the three study regimens (Treatment A - Quinine Sulfate Capsules 324 mg under fasting conditions, Treatment B - Quinine Sulphate Tablets 300 mg under fasting conditions and Treatment C - Quinine Sulfate Capsules 324 mg under fed conditions) in a randomly assigned sequence of dosing periods, each followed by a washout period of 7 days.
Period: Period I
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 9 | 9 | 9
Completed | 9 | 9 | 9
Not Completed | 0 | 0 | 0
Period: Washout Period A
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 9 | 9 | 9
Completed | 9 | 9 | 8 (positive pregnancy test - recorded as an adverse event)
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Period: Period II
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 9 | 9 | 8
Completed | 9 | 9 | 8
Not Completed | 0 | 0 | 0
Period: Washout Period B
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 9 | 9 | 8
Completed | 9 | 9 | 7 (personal reasons)
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Period III
Arm/Group | Treatment Sequence ABC | Treatment Sequence BCA | Treatment Sequence CAB
Started | 9 | 9 | 7
Completed | 9 | 9 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All subjects received each of the three study regimens (Treatment A - Quinine Sulfate Capsules 324 mg under fasting conditions, Treatment B - Quinine Sulphate Tablets 300 mg under fasting conditions and Treatment C - Quinine Sulfate Capsules 324 mg under Fed conditions) in a randomly assigned sequence of dosing periods, each followed by a washout period of 7 days.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.11 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn within one hour prior to dosing (hour 0) and at 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36 and 48 hours after dose administration.
Population: Data for 26 of the 27 subjects were used in the statistical analysis for Treatments A and C. The data for one subject, who dropped from the study prior to period III dosing (Treatment B), was included in the comparison of Treatments A versus C. Treatment A, Dose Adjusted to 300 mg was used to evaluate for dose proportionality.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Treatment A - Quinine Sulfate 324 mg Caps, Fasting Conditions: Each subject received one capsule of Quinine Sulfate 324 mg after an overnight fast of at least 10 hours.
- Treatment A, Dose Adjusted to 300 mg: This group was a statistical adjustment only. Treatment A (Quinine Sulfate 1 x 324 mg Capsule) Dose Adjusted to 300 mg was used to evaluate for dose proportionality.
- Treatment B- Quinine Sulphate 300 mg Tabs, Fasting Conditions: Each subject received one tablet of Quinine Sulphate 300 mg after an overnight fast of at least 10 hours.
- Treatment C - Quinine Sulfate 324 mg Caps, Fed Conditions: Each subject received one capsule of Quinine Sulfate 324 mg thirty minutes after the initiation of a standardized, high-fat breakfast following an overnight fast.
Arm/Group | Treatment A - Quinine Sulfate 324 mg Caps, Fasting Conditions | Treatment A, Dose Adjusted to 300 mg | Treatment B- Quinine Sulphate 300 mg Tabs, Fasting Conditions | Treatment C - Quinine Sulfate 324 mg Caps, Fed Conditions
Number analyzed (Participants) | 26 | 26 | 25 | 26
ng/mL | 2,246.58 (594.69) | 2,080.18 (550.64) | 2,278.46 (547.79) | 2,539.94 (740.19)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Groups:
- Treatment C - Quinine Sulfate 324 mg Caps, Fed Conditions: Each subject received one capsule of Quinine Sulfate 324 mg 30 minutes after the initiation of a standardized, high-fat breakfast following an overnight fast.
Arm/Group | Treatment A - Quinine Sulfate 324 mg Caps, Fasting Conditions | Treatment A, Dose Adjusted to 300 mg | Treatment B- Quinine Sulphate 300 mg Tabs, Fasting Conditions | Treatment C - Quinine Sulfate 324 mg Caps, Fed Conditions
Number analyzed (Participants) | 26 | 26 | 25 | 26
ng-hr/mL | 32,689.35 (8,667.79) | 30,267.96 (8,025.76) | 31,689.32 (9,549.17) | 34,729.00 (11,625.99)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Treatment A - Quinine Sulfate 324 mg Caps, Fasting Conditions | Treatment A, Dose Adjusted to 300 mg | Treatment B- Quinine Sulphate 300 mg Tabs, Fasting Conditions | Treatment C - Quinine Sulfate 324 mg Caps, Fed Conditions
Number analyzed (Participants) | 26 | 26 | 25 | 26
ng-hr/mL | 36,132.35 (11,054.19) | 33,456.04 (10,235.39) | 34,410.28 (11,636.62) | 37,550.81 (14,809.14)

ADVERSE EVENTS:
Groups:
- Treatment A - Quinine Sulfate Capsules 324 mg - Fasting; Treatment B - Quinine Sulphate Tablets 300 mg - Fasting; Treatment C - Quinine Sulfate Capsules 324 mg - Fed: All subjects received each of the three study regimens (Treatment A - Quinine Sulfate Capsules 324 mg under fasting conditions, Treatment B - Quinine Sulphate Tablets 300 mg under fasting conditions and Treatment C - Quinine Sulfate Capsules 324 mg under fed conditions) in a randomly assigned sequence of dosing periods, each followed by a washout period of 7 days.
Arm/Group | Treatment A - Quinine Sulfate Capsules 324 mg - Fasting | Treatment B - Quinine Sulphate Tablets 300 mg - Fasting | Treatment C - Quinine Sulfate Capsules 324 mg - Fed
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 11/26 | 7/25 | 14/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A - Quinine Sulfate Capsules 324 mg - Fasting (N=26) | Treatment B - Quinine Sulphate Tablets 300 mg - Fasting (N=25) | Treatment C - Quinine Sulfate Capsules 324 mg - Fed (N=27)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 3 (3) | 3 (3) | 4 (4)
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
unintended pregnancy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
viral syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5)
syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days